CLINICAL TRIAL: NCT01440361
Title: A Clinical and Mechanistic Proof of Efficacy Study With Belimumab in Chronic Immune Thrombocytopenia (ITP) Patients.
Brief Title: A Study to Investigate Belimumab for the Treatment of Chronic Immune Thrombocytopenia.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was Cancelled Before Active
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 114870
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
MeSH Terms: conditions — Purpura | interventions — belimumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belimumab (Experimental): Reconstituted solution for intravenous infusion
  Interventions: Drug: Belimumab
- Normal saline (Placebo Comparator): Solution for intravenous infusion
  Interventions: Drug: Normal saline placebo

INTERVENTIONS:
Drug: Belimumab — 10 mg /kg given as an intravenous infusion every 4 weeks for 24 weeks (with an additional dose at Week 2)
  Other Names: Benlysta/LymphoStat-B
  Arms: Belimumab
Drug: Normal saline placebo — Placebo given as an intravenous infusion every 4 weeks for 24 weeks (with an additional dose at Week 2)
  Other Names: Saline
  Arms: Normal saline

SUMMARY:
Chronic immune thrombocytopenia (ITP) is a longterm disease in which the blood does not clot normally. This is due to a low number of blood cell fragments called platelets. Platelets clot to seal small cuts or breaks on blood vessel walls and stop bleeding. Normally the immune system makes proteins called antibodies to fight off harmful substances that enter the body. In ITP, the immune system produces antibodies that attack and destroy the body's platelets by mistake.

Patients can suffer from bleeding under the skin, nosebleeds, blood in urine or stools and in very severe cases bleeding in the brain. Patients have an increased frequency of death from bleeding complications compared to normal.

Chronic ITP is fairly rare , with an incidence of 32 new cases/million people each year.

Existing treatments work by lowering the activity of the immune system or directly increasing platelet count. These treatments do not work effectively in all patients and can have side effects. We hope that understanding how belimumab works in ITP will help in the development of future treatments for ITP and other autoimmune diseases.

We will test the safety, blood levels and effects of the study medication in people with chronic ITP. Patients will receive the study medication intravenously (through a needle inserted into a vein) and blood samples will be taken before and on several occasions afterwards.

Up to 40 patients with chronic ITP, aged 18 to 75 will participate. Approximately 11 patients will take dummy medicine instead of the study medicine neither they or their study doctor will know which one they are given. Participants will take up to 57 weeks to finish the study. They'll make 12 outpatient visits.

The study will take place in hospitals in the UK. Other sites in mainland Europe may also be initiated.

A pharmaceutical company, GlaxoSmithKline, is funding the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,18-75 years old
* Chronic ITP for a minimum of 6 months with a platelet count <75,000/uL at screening and a platelet count <75,000/uL 2 to 6 months before screening
* Stable either on no treatment or on a stable dose of corticosteroids (10 milligrams(mg)/day prednisone or prednisone equivalent or less) and/or azathioprine (100mg/day or less) for a minimum of 30 days before screening
* Single QTc <450 milliseconds (msec); or QTc <480 msec in subjects with Bundle Branch Block
* A female subject is eligible to participate if she is not pregnant or nursing and at least one of the following conditions apply: a. Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. b.Child-bearing potential and agrees to use one of the contraception methods listed in the protocol

Exclusion Criteria:

* Diagnosis of ITP is secondary to other conditions
* Treated with any B cell targeted therapy at any time
* Have received any of the following within 364 days prior to Day 0: Abatacept, A biologic investigational agent other than B cell targeted therapy
* Have received any of the following within 180 days prior to Day 0: Intravenous (IV) cyclophosphamide, 3 or more courses of systemic corticosteroids for concomitant conditions
* Have received any of the following within 90 days prior to Day 0: High dose corticosteroid for treatment of ITP, Splenectomy, plasmapheresis
* Have received any of the following within 60 days, 5 half-lives or twice the duration of the biological effect of belimumab before Day 0: A non-biologic investigational agent, any other immunosuppressive/immunomodulatory agent with the exception of azathioprine and corticosteroids, Eltrombopag, romiplostim, any steroid injection
* Have received any of the following within 30 days before Screening: Intravenous immunoglobulin, Corticosteroids greater than 10mg/day (prednisone or prednisone equivalent) or azathioprine more than 100 mg/day, Changes to corticosteroid or azathioprine therapy
* Have received a live vaccine within 30 days before Day 0
* Subject could be at risk of haemorrhage that threatens a vital organ
* History of a major organ transplant or hematopoietic stem cell/marrow transplant
* History of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix
* Required management of infections, as follows: Currently on any suppressive therapy for a chronic infection, Hospitalisation for treatment of infection within 60 days before Day 0, Use of parenteral antibiotics within 60 days before Day 0
* Significant unstable or uncontrolled acute or chronic diseases not due to ITP or planned surgical procedure or a history of any other medical disease, laboratory abnormality, or condition that makes the subject unsuitable for the study
* Positive screening Hepatitis C antibody result or Hepatitis B (HB) infection
* Positive test for Human Immunodeficiency Virus (HIV) antibody at screening or historically
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater or equal to 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
* IgA deficiency (IgA <10mg/dL)
* Abnormal lab results
* Lymphocyte count <500/mm3
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy including a previous anaphylactic reaction to parenteral administration contrast agents, human or murine proteins or monoclonal antibodies
* Evidence of serious suicide risk
* Current drug or alcohol abuse or dependence
* Where participation in the study would result in donation of blood or blood products >500 mL within a 56 day period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Platelet count | Baseline, week 28
  Change in platelet count
Anti-platelet autoantibodies | Baseline, week 28
  Change in anti-platelet autoantibodies

SECONDARY OUTCOMES:
Platelet count (time) | Baseline, week 0, 2, 4, 8, 12, 16, 20, 24, 28
  Time to first response of platelet count increase >20,000/microlitre (μl) from baseline
Platelet count (incidence) | Baseline, week 28
  Incidence of response of platelet count increase >20,000/μL from baseline
Platelet count (incidence of complete response) | Baseline, week 28
  Incidence of complete response as defined by platelet count to >100,000
Platelet count (incidence of doubling) | Baseline, week 28
  Incidence of subjects with ≥2 times baseline platelet count
Vital signs | Baseline, week 0, 2, 4, 8, 12, 16, 20, 24, 28, 40
  Change in vital signs outside normal range
Clinical chemistry and haematology | Baseline, week 2, 4, 8, 12, 16, 20, 24, 28, 40
  Change in clinical chemistry and haematology
Immunogenicity | Baseline, week 12, 28, 40, 52
  Change in immunogenicity
Serum concentrations of belimumab | Baseline, week 2, 8, 24, 28, 40, 52
  Change in serum concentrations of belimumab
Serum and/or platelet bound anti-platelet antibodies | Baseline, week 4, 8, 12, 16, 20, 24, 28, 40, 52
  Change in serum and/or platelet bound anti-platelet antibodies
B cell and T cell sub-populations and B lymphocyte stimulator (BLyS) receptor | Baseline, week 4, 8, 16, 24, 40, 52
  Change in B cell and T cell sub-populations and BLyS receptor
Antigen-specific B cells and T cells | Baseline, week 8, 16, 24, 40
  Change in antigen-specific B cells and T cells
Serum cytokine/chemokine profile | Baseline, week 8, 16, 24, 28, 40
  Change in serum cytokine/chemokine profile
Transcriptome profile | Baseline, week 8, 28
  Change in transcriptome profile
Autoantibody profile | Baseline, week 28
  Change in autoantibody profile

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline